CLINICAL TRIAL: NCT06987656
Title: The Role of Physiotherapy in the Management of Acute Lumbar Spasm in Emergency Departments: A Retrospective Observational Study
Brief Title: Physiotherapy in Emergency Department for Acute Lumbar Spasm
Acronym: PT-ED
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Collaborators: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Veysel Uludag, Lecturer, Duzce University
Other Study IDs: 2024/254
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Acute Low Back Pain; Musculoskeletal Pain; Emergency Care
Keywords: Physiotherapy; Acute Low Back Spasm; Emergency Department; Manual Therapy; Exercise Therapy; Pain Management
MeSH Terms: conditions — Musculoskeletal Pain; Emergencies; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pharmacologic Treatment Only Group: Patients who received standard pharmacologic treatment only, including NSAIDs, muscle relaxants, and analgesics, without any physiotherapy intervention.
  Interventions: Drug: Standard Pharmacologic Treatment
- Pharmacologic + Physiotherapy Group: Patients who received standard pharmacologic treatment along with physiotherapy interventions, including spinal mobilization, electrotherapy (TENS), and individualized exercise programs.
  Interventions: Drug: Standard Pharmacologic Treatment; Other: Physiotherapy Intervention

INTERVENTIONS:
Drug: Standard Pharmacologic Treatment — Standard pharmacologic management including nonsteroidal anti-inflammatory drugs (NSAIDs), muscle relaxants (e.g., thiocolchicoside), and analgesics (e.g., paracetamol, tramadol) for acute lumbar spasm.
Other: Physiotherapy Intervention — Physiotherapy interventions included spinal mobilization (Maitland techniques), myofascial release, transcutaneous electrical nerve stimulation (TENS), and personalized exercise programs, as documented in patient medical records.
  Groups: Pharmacologic + Physiotherapy Group

SUMMARY:
This retrospective observational study aims to evaluate the effectiveness of physiotherapy interventions-such as manual therapy, electrotherapy (TENS), and individualized exercise programs-in managing acute lumbar spasm in patients presenting to the emergency department. By analyzing medical records from January to June 2024 at Düzce University Faculty of Medicine, the study will compare outcomes between patients receiving only pharmacological treatment and those receiving additional physiotherapy. Primary outcomes include changes in pain levels (measured by Visual Analog Scale), medication usage, patient satisfaction, and re-admission rates within an 8-week follow-up period. The findings aim to inform the integration of physiotherapy into emergency care protocols for acute lumbar spasm.

DETAILED DESCRIPTION:
This retrospective observational study investigates the role of physiotherapy in managing acute lumbar spasm in emergency department settings. The study will review medical records of 100 patients aged 18 to 65 who presented to Düzce University Faculty of Medicine Emergency Department between January and June 2024 with non-specific acute low back spasm.

Patients will be divided into two groups based on documented treatment: (1) those receiving pharmacological treatment only, and (2) those receiving both pharmacological and physiotherapy interventions. Physiotherapy interventions include spinal mobilization, myofascial release, TENS (Transcutaneous Electrical Nerve Stimulation), and individualized exercise protocols.

Primary outcomes include changes in pain intensity (measured by Visual Analog Scale), medication consumption, re-admission rates within 8 weeks, and overall patient satisfaction. The study also incorporates a cost analysis based on national reimbursement tariffs (SUT) to evaluate the financial impact of integrating physiotherapy into emergency care.

This study does not involve any direct intervention, and data are collected exclusively from existing electronic health records. Ethical approval has been obtained. The findings are expected to guide future protocols involving the integration of physiotherapy into emergency departments in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 65 years
* Presented to the emergency department with non-specific acute lumbar spasm
* No serious pathology on initial evaluation (e.g., infection, malignancy, fracture)
* No contraindications to physiotherapy or physical activity
* Agreed to participate in the study and signed the informed consent (if applicable in prospective cases)

Exclusion Criteria:

* History of chronic low back pain
* Presence of neurological deficits (e.g., paresis, paralysis)
* Diagnosed with serious medical conditions such as infection, malignancy, or spondylodiscitis
* Pregnancy or contraindications related to reproductive health
* History of spinal surgery within the past year
* Cognitive or physical impairments limiting treatment participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult patients aged 18 to 65 who are admitted to the Emergency Department of Düzce University Faculty of Medicine between June 1, 2025, and December 25, 2025, with a diagnosis of non-specific acute lumbar spasm. The study will retrospectively analyze data from electronic medical records to evaluate physiotherapy and pharmacologic treatment outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity Measured by Visual Analog Scale (VAS) From Admission to Discharge | VAS score (0-10 scale)
  At Emergency Department Admission and at Time of Discharge (up to 12 hours)

SECONDARY OUTCOMES:
Level of Patient Satisfaction Recorded at Discharge | At Discharge (within 12 hours of Emergency Department Admission)
  Patient satisfaction levels will be assessed using standardized satisfaction forms documented in the electronic medical record system at the time of discharge. Data will be extracted retrospectively and categorized as satisfied, neutral, or dissatisfied, based on the available hospital documentation.

CONTACTS AND LOCATIONS:
Locations (1):
- Duzce University, Düzce, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the retrospective nature of the study and the use of sensitive patient information obtained from electronic medical records. The study does not include prior consent for data sharing, and confidentiality regulations prohibit the distribution of such data.

REFERENCES:
- [Derived] Uludag V, Tekin RT, Bogan M, Senguldur E, Demir MC. Integrating physiotherapy into the emergency department for acute low back spasm: a retrospective comparative study. Physiother Theory Pract. 2026 Jan 30:1-10. doi: 10.1080/09593985.2026.2624519. Online ahead of print. PMID 41614542